CLINICAL TRIAL: NCT01740011
Title: A Prospective Randomized Trial on Comparison of Standard- Carbon Dioxide Pressure Pneumoperitoneum Insufflators Versus AirSeal
Brief Title: Prospective Randomized Trial on Comparison of Standard- Carbon Dioxide Pressure Pneumoperitoneum Insufflators Versus AirSeal
Acronym: AirSeal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Krankenhaus Barmherzige Schwestern Linz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AT-1112-RL
Record Dates: First submitted 2012-11-23; First posted 2012-12-04 (Estimated); Last update posted 2014-09-08 (Estimated); Status verified 2014-01

CONDITIONS: Colorectal Disorders; Hernia; Incidence for Cholecystectomy
MeSH Terms: conditions — Hernia | interventions — Laparoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Experimental): Laparoscopic surgery with AirSeal CO2 pressure insufflation
  Interventions: Procedure: Laparoscopic surgery
- Group S (Active Comparator): Laparoscopic surgery with standard CO2 pressure insufflation
  Interventions: Procedure: Laparoscopic surgery

INTERVENTIONS:
Procedure: Laparoscopic surgery

SUMMARY:
The primary objective of the present trial is to investigate, the mean operative time and to study the frequency and intensity of postoperative shoulder tip pain in patients undergoing laparoscopic surgery, i.e. cholecystectomy, colorectal surgery, hernia repair with AirSeal® compared with standard pressure CO2 insufflation systems. The primary hypothesis is that patients operated with AirSeal® have a shorter mean operative time and decreased frequency and intensity of postoperative shoulder tip pain compared with patients undergoing surgery with standard pressure CO2 insufflation systems.

It is the secondary objective of the trial to evaluate immunologic and anaesthesiological aspects of laparoscopic cholecystectomy, colorectal surgery and laparoscopic hernia repair by observing the immune responses and volume of mechanical ventilation of the two groups through measuring various immunologic factors and ventilation volume/CO2 elimination volume. Surgical side effects will also be measured as secondary objective.

ELIGIBILITY:
Inclusion Criteria:

* Patients recruited for laparoscopic surgery i.e. cholecystectomy, colorectal surgery, hernia repair
* Written informed consent
* ≥ 18 years of age

Exclusion Criteria:

* Patients with known immunological dysfunction (advanced liver disease, HIV, hepatitis C virus infection), drug addiction
* ≤18 years of age
* Pregnancy and lactation
* Previous extensive abdominal surgery
* Acute surgical intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Estimated)
Dates: Start 2013-01; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
time of surgery | one year
  Time of surgery, expressed in minutes from the time of incising to suturing the skin.
shoulder pain | one year
  Postoperative shoulder tip pain assessed by the Visual Analogue Scale of Pain (VAS scale).

SECONDARY OUTCOMES:
Immunological aspects | one year
  Examine changes in the concentration of certain cytokines and angiogenic factors serum levels in the early postoperative period after laparoscopic surgery procedures performed with AirSeal® versus standard- pressure CO2 pneumoperitoneum.
postoperative complications | one year
  Haemorrhage, Wound infections, Intra-abdominal abscess, Anastomotic leakage, Deep vein thrombosis, Pulmonary embolism

OTHER OUTCOMES:
Anaesthesiological aspects | one year
  Examine intraoperative changes in ventilation volume, acid-base balance and CO2 elimination in patients undergoing laparoscopic surgery procedures performed with AirSeal® versus standard- pressure CO2 pneumoperitoneum.

CONTACTS AND LOCATIONS:
Overall Officials: Ruzica-Rosalia Luketina, MD, Principal Investigator — Krankenhaus Barmherzige Schwestern Linz
Locations (1):
- Krankenhaus der Barmherzigen Schwestern Linz, Linz, Upper Austria, Austria

REFERENCES:
- [Derived] Gallioli A, De Lorenzis E, Lievore E, Boeri L, Colombo L, Fontana M, Breda A, Montanari E, Albo G. The Effect of CO2 Pressure and Flow Variation on Carbon Particles Spread During Pneumoperitoneum: An Experimental Study. J Endourol. 2022 Jun;36(6):807-813. doi: 10.1089/end.2021.0336. Epub 2022 May 17. PMID 34779236
- [Derived] Luketina R, Luketina TLH, Antoniou SA, Kohler G, Konneker S, Manzenreiter L, Wundsam H, Koch OO, Knauer M, Emmanuel K. Prospective randomized controlled trial on comparison of standard CO2 pressure pneumoperitoneum insufflator versus AirSeal(R). Surg Endosc. 2021 Jul;35(7):3670-3678. doi: 10.1007/s00464-020-07846-4. Epub 2020 Aug 7. PMID 32767145
- [Derived] Luketina RR, Knauer M, Kohler G, Koch OO, Strasser K, Egger M, Emmanuel K. Comparison of a standard CO(2) pressure pneumoperitoneum insufflator versus AirSeal: study protocol of a randomized controlled trial. Trials. 2014 Jun 20;15:239. doi: 10.1186/1745-6215-15-239. PMID 24950720
- See also: Investigator related informations — http://www.bhs.at